CLINICAL TRIAL: NCT03117296
Title: Physical Therapy and Occupational Therapy After Transcatheter Aortic Valve Replacement
Acronym: PTOTtAVR
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Principal Investigator, Adele Myszenski, Supervisor, Physical Therapist, Henry Ford Health System
Other Study IDs: 10437
Record Dates: First submitted 2017-04-07; First posted 2017-04-17 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-04

CONDITIONS: Transcatheter Aortic Valve Implantation
Keywords: physical therapy; occupational therapy; tAVR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post procedure routine PT and or OT: Routine PT and or OT
  Interventions: Other: Routine PT or OT
- Post Procedure PT and OT pathway: Post procedure day zero nursing mobilization; post procedure day one PT and OT assessment and intervention, daily PT and OT intervention
  Interventions: Other: Post procedure daily PT and OT; Other: PT post procedure; Other: OT post procedure

INTERVENTIONS:
Other: Post procedure daily PT and OT — PT evaluation and treatment on post procedure day zero: Nurses mobility patient using egress testing one time
  Groups: Post Procedure PT and OT pathway
Other: PT post procedure — post procedure day one: PT and OT assessment, education and intervention.
  Groups: Post Procedure PT and OT pathway
Other: OT post procedure — PT and OT Daily until goals met or patient discharge.
  Groups: Post Procedure PT and OT pathway
Other: Routine PT or OT — Routine PT or OT consulted by physician when identified discharge disposition of home
  Groups: Post procedure routine PT and or OT

SUMMARY:
Implementation of Physical Therapy (PT) and Occupational Therapy (OT) pathway (initiation of services on Post procedure day #1 and continued daily with focus on education and activity progression) for all patients undergoing a transcatheter aortic value repair procedure began on December 2, 2014. Retrospective data was collected from The Society of Thoracic Surgeons/American College of Cardiology Transcatheter Aortic Valve Replacement Procedures (STS/ACC TVT, trademark) Registry - National database for Transcatherter Aortic Valve Replacement Procedures and included subjects from March 2012 through July 31, 2015. Patients included: s/p tAVR via transfemoral catheter approach, with or without minor intra or post procedure events (GI bleeds, minor access bleeds, afib, etc); Exclusions: Major events including stroke, pacemaker placement, other cardiovascular (CV) repair or surgery required, etc). Future data analysis will extend subjects to December 31, 2015 and annually.

DETAILED DESCRIPTION:
Rationale: Frequency of transcatheter and other structural heart procedures increased dramatically from 2012 to 2014 and is trending even higher for 2015. Procedures increased from 15 in 2012 to 50 cases in 2013 (233% increase) and to 70 cases in 2014 (40% increase from 2013 to 2014.) -- PT and OT identified a gap in consults and need for specific education targeted for a new surgery population (tAVR) without sternotomy. Often consults were placed on day of discharge to rehab facility or not at all. -- Structural Heart division of CV institute identified increased length of stay (LOS) and decreased activity of their patients in the hospital. -- No literature on this subject found via Henry Ford Hospital Sladen Library PubMed literature review

Aim: • Create a standardized pathway for new transcatheter aortic valve replacement patients in the Structural Heart Division (SHD)

* Improve patient outcomes including increasing the percentage of patients returning to home rather than a rehab facility destination at discharge
* Decrease length of stay

Implementation:

* Plan: PT and OT identified a gap in consults and need for specific education targeted at a new surgeries population (tAVR); Structural Heart division of CV institute identified an increase LOS and decreased activity of their patients in the hospital. In October 2014 planning began to introduce a SHD tAVR pathway that would include post procedure day number 0 nursing requirements and training, post procedure day number 1-3 PT and OT assessment and interventions.
* Do: Implemented pathway in November 2014.
* Check: Order set revision; Patient handouts ; Cardiac Rehab; Weekend criteria; staff training
* Act: February 2015, order sets in place, patient handouts finalized and full pathway finalized for post op tAVR patients.
* Continued checks identified additional SHD procedures and team determined that Mitral Clips and LARIATs were not criteria for tAVR pathway but would receive routine PT and OT consults.

Intervention: • Added PT and OT to Structural Heart Order Set.

* PT and OT assessments completed on post procedure day number day 1.
* PT and OT follow up treatments post procedure day number 2, 3 and beyond as appropriate.
* Patient education handouts individualized for patient population
* Pre-op education handouts individualized for patient population

Outcome measures: Hospital Length of stay, discharge disposition. Data Analysis: Chi-square tests are used to compare proportions between groups, while Wilcoxon two-sample tests are used to compare distributions of continuous variables between groups. This nonparametric test was chosen due to non-Gaussian distribution of the continuous outcomes within groups. Statistical significance was set at p<0.05. All analyses were performed using SAS 9.4 (SAS Institute Inc, Cary, North Carolina, USA).

ELIGIBILITY:
Inclusion Criteria:

* admission to henry ford hospital after March 1, 2012
* status post transcatheter aortic valve replacement via transfemoral catheter approach, with or without minor intra or post procedure events (GI bleeds, minor access bleeds, afib, etc)

Exclusion Criteria:

* Occurrence of major events including stroke, pacemaker placement, other CV repair or surgery required, etc)
* procedure via appropriate other than femoral access (transapical, transcaval)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive population sample of patients at Henry Ford Hospital, Detroit, Michigan undergoing transcatheter aortic valve replacement via femoral access in cath lab from March 2012 to present.
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Myszenski, MPT, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
IRB was closed March 08-2021 and no plans to share data from this preliminary study

REFERENCES:
- [Background] Babaliaros V, Devireddy C, Lerakis S, Leonardi R, Iturra SA, Mavromatis K, Leshnower BG, Guyton RA, Kanitkar M, Keegan P, Simone A, Stewart JP, Ghasemzadeh N, Block P, Thourani VH. Comparison of transfemoral transcatheter aortic valve replacement performed in the catheterization laboratory (minimalist approach) versus hybrid operating room (standard approach): outcomes and cost analysis. JACC Cardiovasc Interv. 2014 Aug;7(8):898-904. doi: 10.1016/j.jcin.2014.04.005. Epub 2014 Jul 30. PMID 25086843
- [Background] Marcantuono R, Gutsche J, Burke-Julien M, Anwaruddin S, Augoustides JG, Jones D, Mangino-Blanchard L, Hoke N, Houseman S, Li R, Patel P, Stetson R, Walsh E, Szeto WY, Herrmann HC. Rationale, development, implementation, and initial results of a fast track protocol for transfemoral transcatheter aortic valve replacement (TAVR). Catheter Cardiovasc Interv. 2015 Mar;85(4):648-54. doi: 10.1002/ccd.25749. Epub 2014 Nov 29. PMID 25413312
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective study of patients whom received a tAVR procedure via transfemoral catheter percutaneous access site in the catheterization laboratory at HFH from March 1, 2012, to December 31, 2015. Exclusion criteria included access sites other than femoral, the occurrence of major events.
Pre-assignment Details: Patients excluded from database included those with an access sites other than femoral, the occurrence of major events including death, stroke, myocardial infarction (MI), additional cardiac or vascular surgery, electrophysiological monitoring, pacemaker placement, atrial fibrillation, other car-diovascular repair or surgery required, gastrointestinal bleeds, hematoma or access bleeds, or complications
Groups:
- Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation: Routine PT and or OT
  Routine PT or OT: Routine PT or OT consulted by physician when identified discharge disposition of home
- Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation: Post procedure day zero nursing mobilization; post procedure day one PT and OT assessment and intervention, daily PT and OT intervention
  Post procedure daily PT and OT: PT evaluation and treatment on post procedure day zero: Nurses mobility patient using egress testing one time
  PT post procedure: post procedure day one: PT and OT assessment, education and intervention.
  OT post procedure: PT and OT Daily until goals met or patient discharge.
Period: Overall Study
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Started | 74 | 115
Completed | 74 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation | Total
Number analyzed (Participants) | 74 | 115 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.5 (11.2) | 81.6 (8.4) | 80.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 47 | 79
  Male | 42 | 68 | 110
Region of Enrollment [Number; unit: participants]
  United States | 74 | 115 | 189
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (6.2) | 28.4 (6.1) | 28.4 (6.2)
Society of Thoracic Surgeons Risk Score [Mean (Standard Deviation); unit: Percentage] — The Society of Thoracic Surgeons adult cardiac surgery risk model calculates patient's risk of mortality & morbidities for the most common cardiac surgeries; estimates should be considered as only 1 of several sources of information in decision-making and patient counseling. The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database.1 In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk. J INVASIVE CARDIOL 2017;29(3):109-114
  Percentage | 8.5 (8.5) | 7.0 (4.6) | 7.75 (6.6)
Valve Sheath Delivery Size [Mean (Standard Deviation); unit: milimeter diameter of tAVR device] — Society of Thoracic Surgeons Registry records the size of the catheter used during the tAVR procedure. Sizes range from 17.8 to 30.1. The latest generation of TAVR devices have incorporated features to reduce the delivery catheter profile, facilitate deployment, and enable repositioning and retrieval capability, with the aim of obtaining the desired position and reducing TAVR-related complications. https://citoday.com/pdfs/cit0317_F5_Barbanti.pdf This variable was initially an important way to control for the fact that over time from 2013 to 2015, smaller sizes can reduce complications.
  milimeter diameter of tAVR device | 18.1 (4.2) | 19.3 (3.8) | 18.7 (4)

OUTCOME MEASURES:

1. Primary Outcome: Post Procedure Hospital Length of Stay
Description: From date of procedure until date of hospital discharge, assessed up to 50 days.
Time Frame: at discharge
Population: Adults admitted to Henry Ford Hospital and received a transcatheter aortic valve replacement via femoral access site and free from major events or complications.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Number analyzed (Participants) | 74 | 115
days | 4.8 (2.9) | 3.5 (4.0)

2. Primary Outcome: Total Hospital Length of Stay
Description: Days from Hospital admission to Hospital Discharge
Time Frame: at discharge
Population: Adults admitted to HFH and s/p tAVR via femoral site, free from events or complications
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Number analyzed (Participants) | 74 | 115
days | 6.9 (5.4) | 4.5 (5.4)
Statistical Analysis 1: Comparison: Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation vs Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation; Univariate 2-group comparisons were performed using χ2 and Fisher's exact tests (when expected cell counts are <5) for categorical variables, using 2-group t tests and Wilcoxon rank-sum tests (when normality distributions were violated) for continuous variables. Statistical significance was set at P < .05. All analyses were performed using SAS 9.4 (SAS Institute, Cary, North Carolina); Test type: Other; p < 0.01, Fisher Exact; Rank-Sum = .05

3. Secondary Outcome: Discharge Disposition, Home
Description: Discharge destination at discharge. Home includes those discharge home, Home with assistance or Home with Home care.
Time Frame: on day of hospital discharge
Population: Adults admit to HFH and s/p TAVR via femoral access, free from events or complications
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Number analyzed (Participants) | 74 | 115
Participants | 57 | 99

4. Secondary Outcome: Discharge Destination, Rehab Facility
Description: At hospital discharge, did the patient return Home or were they discharged to a post-acute care Rehab Facility
Time Frame: on day of hospital discharge
Population: Adults admit to HFH and s/p tavr via femoral, no events or complications
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Number analyzed (Participants) | 74 | 115
Participants | 17 | 16

ADVERSE EVENTS:
Time Frame: This was a retrospective study.
Description: This was a retrospective study.
Arm/Group | Control Group (TAVR 3/1/12-11/1/14) Pre PT OT Pathway Implementation | Intervention Group (TAVR 11/2/14-12/31/15) Post PT OT Pathway Implementation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One hospital in one area. Low subject number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes